CLINICAL TRIAL: NCT03409406
Title: Using Mobile Health Technology to Optimize Communication Outcomes for South African Children With Developmental Disabilities
Brief Title: Communication Outcomes for South African Children With Developmental Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: University of Pretoria (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Maryann Romski, Regents Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21DC015225 (NIH); R21DC015225 (NIH)
Record Dates: First submitted 2018-01-10; First posted 2018-01-24 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Developmental Disability
Keywords: developmental disability; speech and language disorder; mobile health technology; parent training; communication intervention
MeSH Terms: conditions — Developmental Disabilities; Speech; Language Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiver Intervention + ST Intervention (Experimental): Parents/caregivers receive web-based tablet protocol containing sequenced communication information for working with their child at home in addition to the Standard of Care Intervention.
  Interventions: Behavioral: Caregiver Intervention; Behavioral: ST Intervention
- ST Intervention (Active Comparator): This intervention is the once monthly standard of care intervention 30-minutes speech therapy (ST) session that the child receives at the hospital.
  Interventions: Behavioral: ST Intervention

INTERVENTIONS:
Behavioral: Caregiver Intervention — This intervention is a 3-month (or 12 weeks) sequenced mobile health intervention provided to the parent/caregiver to use at home with the child. It supplements the 30 minute speech and language therapy session provided to the child at the hospital once a month
  Arms: Caregiver Intervention + ST Intervention
Behavioral: ST Intervention — This intervention is the 30 minute speech and language therapy session provided to the child at the hospital once a month for three months.

SUMMARY:
The goal is to remediate speech and language disorders early in the lives of South African children with significant developmental disorders (DD) by enhancing the health care service delivery system to better serve families across diverse backgrounds. This study assesses a new hybrid intervention to promote better communication skills for both the child and caregiver. The hybrid intervention includes a mobile health technology (MHT) web-based tablet protocol that assists parents/caregivers in communicating with their children on a daily basis at home over a 12-week period in addition to the current standard of care intervention, a 30-minute speech-language therapy session at the secondary/tertiary hospitals once a month. The hybrid intervention adds to the child's monthly therapy session by providing parents/caregivers with instruction about communication with their children via a sequenced web-based tablet protocol across a 12 week time period and face-to-face monthly follow-up at the hospital where the child receives therapy. Fifty parent/caregiver-child pairs (25 per group) will be assigned to either the hybrid intervention or the standard of care intervention. Child receptive and expressive language skills, child and parent/caregiver communication interactions and parent/caregiver and speech therapist satisfaction with child communication will be measured prior to the intervention and then again at the end of the 12-week period. The effects of the hybrid intervention and standard of care intervention on child communication skills, caregiver perception and satisfaction and speech therapist perception and satisfaction will be measured. The expectation is that the new MHT enhanced hybrid intervention program that is applicable and deliverable in culturally and linguistically diverse settings will enhance the child's receptive and expressive communication skills and result in greater parent/caregiver and speech therapist satisfaction related to the child. The impact includes enhanced health care service delivery to South African children with DD and their families so as to better serve the children with DD by remediating speech and language disorders on a daily basis.

DETAILED DESCRIPTION:
Children with developmental disorders (DD), such as intellectual disability, autism spectrum disorder, cerebral palsy and other genetic disorders, that affect development and functioning, are at extremely high risk for developing speech and language disorders secondary to their primary condition. Speech and language disorders result in great difficulty communicating with others including primary caregivers, families, peers, and health care providers. These disorders and resulting communication difficulties negatively impact the child's growth, quality of life, long-term development, and later employment reducing the child's ability to contribute to society. Critical barriers to progress in intervention to remediate these difficulties, in countries such as South Africa, are that (1) children with DD and their families often live far from secondary and tertiary hospitals where speech and language intervention services are provided, (2) the families have diverse linguistic backgrounds and (3) health care providers have overwhelmingly large caseloads that result in reduced access to interventions. These issues impact the delivery of services to children with DD, whose speech, language and communication skills are significantly delayed and negatively affect the children's ability to participate, develop and learn at home and in the community.

This clinical trial will improve scientific knowledge about the effects of communication intervention on children's development by enhancing health care service delivery via mobile health technology (MHT) to South African children with DD and differing language backgrounds and their families by remediating speech and language disorders. This project will provide empirical data about the intervention approach and child and caregiver communication outcomes across languages that can be used as the basis for improvement of existing intervention programs. Using a web-based tablet intervention to assist caregivers in communicating with their children on a daily basis in the natural environment providing increased intervention opportunities for the child; 2) manipulate the interventions to promote and improve communication skills for both the child and caregiver; and 3) improve caregiver and speech-language pathologist satisfaction with child communication intervention;

The monthly interventions that the children currently receive at secondary/tertiary hospitals will be supplemented by providing caregivers with improved and enhanced training about communication with their children. This training will be coupled with regular ongoing information via MHT when they return home. This intervention strategy will provide empirical evidence for the role of communication intervention enhanced by MHT in assisting caregivers to implement communication strategies at home on a regular basis.

When the proposed aims are achieved, South African health care service delivery related to speech and language disorders for children with DD will have an empirically-tested strategy for caregiver enhanced intervention of speech and language disorders that can be delivered via MHT in local communities in the family's language. This outcome is in line with the mission and needs of the Fogarty International Center (FIC) and National Institute of Deafness and Other Communication Disorders (NIDCD). Our project will provide a novel approach to health care service delivery that will allow for enhanced collaboration between the speech-language pathologist and the caregiver.The advantages of the program includes the ability to implement communication interventions for children with DD in more locations and provide these children with more frequent communication intervention services through the use of MHT.

Approach The approach is to test the hypothesis that children with DD and their primary caregivers who receive a communication intervention enhanced by MHT will have more developed communication interaction skills than children who receive the standard secondary/tertiary care intervention. The interventions will be manipulated and measure child and caregiver communication interactions and caregiver and speech-language pathologist satisfaction with child communication intervention.

Design: A randomized control design in which children identified with speech and language disorders will be randomly assigned to either an experimental or standard of care group will be employed. All children will be assessed on the assessment battery prior to beginning their participation and again at the end of the intervention. The Experimental group will receive the MHT-enhanced intervention in addition to the standard monthly speech and language intervention provided by the clinic and the standard of care group will continue to receive only the standard communication intervention for a 12-week-period. After that time, the children will be re-assessed to determine changes in communication skills.

Participants. Young children with DD between the ages of 3-6 years who are receiving speech and language services in secondary/tertiary hospitals and their primary caregivers will be participants in this study. Fifty children and their primary caregivers (n = 25 Experimental Group, n = 25 Standard of Care Group) will be recruited. The caregiver will be asked if they are interested in participating in the study. If they agree to participate and complete the informed consent,the children will be assessed in their home language using the communication assessment battery (CAB) developed during the previous Fogarty grant. The child and caregiver will be randomly assigned to the experimental or standard of care groups. Given the previous experience, the expectation is that the overwhelming majority of the young children with DD that are identified will have significant speech and language impairments in their native language. That is, they will primarily be speaking in single words and phrases with varying levels of speech comprehension skills and somewhat impaired speech intelligibility. Some of the children will not be speaking at all. Thus, the focus of the intervention will typically be at the earlier stages of communication development.

Intervention. The supplemental intervention will consist of a primary caregiver communication training program that will be delivered by the research staff in a local primary care setting. It will begin with at least two 1-hr sessions in the caregiver's language including information about communication development and interaction strategies for communicating with the child and practice on the use of the web-based tablet protocol. The caregiver communication training program will use video examples of communication interactions, short lectures/discussions, written materials as appropriate, and role playing activities to teach the caregiver about communicating with the child. It will include segments on: 1) characterizing the individual child's receptive and expressive language and communication skills (based on the CAB assessment), 2) identifying communication challenges the caregiver perceives, 3) identifying initial environments and routines for communication at home, and 4) using the tablet intervention to support in home communication with the child including practice 4 days per week across routines. Principles of adult learning (i.e., role playing, providing opportunities for hands-on practice, creating a open atmosphere in which caregivers can ask questions, including a refresher on the previous session's information will be included. This approach will enable the caregivers to prepare for implementing the tablet protocol at home with the child. The training feedback will use a consistent format beginning with asking for caregiver thoughts and perspective about the session, followed by positive feedback and areas of needed support and concluding with a summary. Once the caregiver returns home with the child, they will use the tablet protocol in a sequential fashion to communicate with their child during activities each week. The caregiver can also use the tablet to obtain refreshers on communication interaction strategies and how to employ them, ask questions and seek guidance. The tablet will also collect data about how the caregiver is using it over time. The clinician will have a face-to-face check-in with the caregiver during the monthly treatment session at the hospital clinic. This check in will provide an opportunity to touch base and gain a sample of how the caregiver child interaction is progressing.

Measures. All children will be assessed using the Communication Assessment Battery (CAB) at each time point throughout their participation. The CAB will be supplemented with 1) general information (medical history and etiology/diagnosis, socio-economic status, family composition, as well as assessment/intervention history including types of intervention) and 2) the adapted Mullen Early Learning Scales in the child's home language to gain a measure of general development from birth up to 68 months of age. This scale measures skills in five areas: Gross Motor, Visual Reception, Fine Motor, Expressive Language, and Receptive Language.

CAB. Standardized and observational measures will be employed. The receptive and expressive language sub-scales of the Mullen will be used to gain data about the child's language skills. The 10 minute caregiver-child interaction sample will permit an examination of the communication interaction skills of the child and the caregiver. The communication interaction sample will be transcribed using the Systematic Analyses of Language Transcripts (SALT) and then employ previously developed coding schemes to measure conversational interaction skills for the child and the caregiver (e.g., turn taking, lexical diversity, mean length of utterance in words). With respect to caregiver perception of child communication, the South African Caregiver Perception of Language Development (SA-CPOLD) which provides a specific measure of the caregiver's perception/satisfaction of issues related to the child's communication development will be administered. It is a paper and pencil survey. On each item, the caregiver responds to a statement using a Likert scale of 1 (strongly disagree) to 5 (strongly agree). A low score (15) would suggest a relatively negative perception of the child's communication development while a high score (45) would suggest a relatively positive perception of the child's communication development. A comparable questionnaire will be developed to assess the speech-language pathologists satisfaction with the MHT-enhanced intervention.

Measures of Web-based tablet protocol use by caregivers. Each week data will be collected from the caregiver on the tablet about their perception of the week's activities.

Data Analyses. In order to answer the research questions associated with Aim 2 of the study, a 2 (intervention group) X 2 (assessment time point) mixed repeated measures ANOVA will be conducted. Power analyses indicate that with an alpha of .05 and power of .80, a total sample size of 50 participants (25 participants in each group) will be needed to detect a moderate effect size.

ELIGIBILITY:
Inclusion Criteria:

* child diagnosis of severe developmental delay with beginning communication skills;
* child receiving monthly speech and language therapy in secondary/tertiary care hospital in northern South Africa

Exclusion Criteria:

* None

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Receptive Language Skills | 3 months
  Receptive Language sub-scale of the Mullen Scales of Early Learning (MSEL) in child's native language. It provides a score in months of age.
Expressive Language Skills | 3 months
  Expressive Language sub-scale of the Mullen Scales of Early Learning (MSEL) in child's native language. It provides a score in months of age.

SECONDARY OUTCOMES:
Caregiver Child Interaction Measures | 3 months
  The 10-minute video interaction between the caregiver and child will be transcribed and mean length of utterance will be calculated for parent and child
SA CPOLD | 3 months
  South African Caregiver Perception of Language Development Measure consists of 15 statements that the caregiver rates on a 1-5 Likert scale. It provides a score of from a low score of 15 to a high score of 45.
SA SLPPOLD | 3 months
  South African Speech Language Pathologist Perception of Language Development Measure will consist of 15 statements that the speech therapist rates on a 1-5 Likert scale. It provides a score of from a low score of 15 to a high score of 45.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Bornman, Ph.D., Principal Investigator — University of Pretoria, South Africa; MaryAnn Romski, Ph.D., Principal Investigator — Georgia State University
Locations (1):
- Center for Augmentative and Alternative Communication, Pretoria, Guatung, South Africa

IPD SHARING:
Plan to Share IPD: Undecided